CLINICAL TRIAL: NCT03217617
Title: Gene Therapy for X-linked Severe Combined Immunodeficiency (SCID-X1) Via Direct Intravenous Injection of Lentiviral Vector (Ivlv-X1)
Brief Title: SCID-X1 Gene Therapy Via Intravenous Lentiviral (Ivlv-X1) Injection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17014
Record Dates: First submitted 2017-07-03; First posted 2017-07-14 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: SCID, X-Linked
Keywords: SCID-X1; lentiviral vector; intravenous gene transfer
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): In vivo LV gene transfer to treat SCID-X1
  Interventions: Biological: Direct intravenous injection of ivlv-X1 lentiviral vector

INTERVENTIONS:
Biological: Direct intravenous injection of ivlv-X1 lentiviral vector — ivlv-X1 LV intravenous injection at a dose of ~1x10e9/kg body weight.

SUMMARY:
This is a Phase I/II gene therapy trial treating X-linked severe combined immunodeficiency (SCID-X1) using a self-inactivating lentiviral vector (ivlv-X1) to functionally correct the genetic defect. The primary objectives are to evaluate the safety and efficacy of the direct intravenous lentiviral gene transfer protocol.

DETAILED DESCRIPTION:
X-linked severe combined immunodeficiency (SCID-X1) is a genetic disorder caused by defect in the common cytokine receptor chain, normally on the surface of lymphocytes. Individuals with SCID-X1 lack the normal development of a functional immune system and so have difficulty fighting infections, which may lead to chronic or severe illness and death. X-SCID patients are normally rescued by a bone marrow transplant from a healthy donor. This trial aims to treat SCID-X1 using a self-inactivating lentiviral vector (LV) carrying a functional gene to correct the genetic defect. By direct intravenous (iv) injection of the LV (ivlv-X1) to modify immune cells in the body, this treatment may establish normal healthy immune cells and overcome the immunodeficiency.

The primary objectives are to evaluate the safety of the self-inactivating ivlv-X1-LV, the in vivo gene transfer protocol and the efficacy of immune reconstitution in patients overcoming frequent infections present at the time of treatment, assessment of iv LV gene transfer efficiency, and finally the long-term correction of immunodeficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SCID-X1 based on:

   * A proven mutation in the common interleukin-2 receptor gamma chain gene as defined by direct sequencing of patient DNA.
   * T-cell immune deficiency defined as one or more of the following: CD3+ autologous T cells < 300/ul, or less than 50% of normal value for in vitro mitogen stimulation, or absent proliferation in vitro to antigen stimulation.
2. No available HLA identical related donor.
3. With severe infections, including but not limited to: pneumonitis; protracted diarrhea requiring total parenteral nutrition; infection with herpes viruses or adenovirus; disseminated BCG infection.
4. No cytogenetic abnormalities (medullary karyotype) and no detection of main rearrangements associated with acute leukemia.
5. No prior allogeneic stem cell transplantation.
6. Life expectancy ≥ 3 months.
7. Documented to be negative for HIV infection.
8. Written, informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

1. No available molecular diagnosis confirming SCID-X1.
2. Existence of an available HLA-identical related donor.
3. Diagnosis of active malignant disease other than EBV-associated lymphoproliferative disease.
4. Current treatment with any chemotherapeutic agent (becomes eligible if not on treatment for at least 1 month).
5. Patients with evidence of infection with HIV-1 or 2.
6. Presence of a medical condition indicating that survival will be less than 4 weeks such as the requirement for mechanical ventilation, severe failure of a major organ system, or evidence of a serious, progressive infection that is refractory to medical treatment.
7. Current treatment with any immunosuppressive agent, excluding corticosteroids.
8. Patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 1 Month to 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
Overall immune reconstitution | 1 year
  T and B cell recovery
Change of infection status | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Ph.D, Principal Investigator — Shenzhen Geno-Immune Medical Institute; Qiyong Zhu, MD, Study Director — Guilin Hospital of Chinese Traditional and Western Medicine
Locations (2):
- China (2):
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Guilin Hospital of Chinese Traditional and Western Medicine, Guilin, Guangxi

IPD SHARING:
Plan to Share IPD: No